CLINICAL TRIAL: NCT04892134
Title: Evaluation of Clinical, Morphologic and Biochemical Markers in Multiple Sclerosis - MarkMS
Brief Title: Evaluation of Clinical, Morphologic and Biochemical Markers in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: MarkMS
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: biomarker; progression; MRI; cognition
MeSH Terms: conditions — Multiple Sclerosis; Disease Progression | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, peripheral blood mononuclear cells, DNA, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample — 40-50 ml of blood is taken

SUMMARY:
By combining clinical, morphological and biochemical markers a better understanding of the formation and progression of multiple sclerosis (MS) should be obtained

DETAILED DESCRIPTION:
The current study aims to comprehensively investigate the individual clinical, morphological and biochemical aspects of MS in order to elucidate underlying mechanisms leading to disease progression. This shall ultimately serve to identify imaging and biochemical markers, which may support clinical management of persons with MS (pwMS). The following markers will be assessed: demographics (age, sex), clinical (EDSS at baseline, disease duration); neuropsychological (SDMT (Symbol Digit Modalities Test) score); MRI (Magnetic Resonance Imaging) (lesion load, atrophy); Biochemical markers analyzed in cerebrospinal fluid (CSF), blood, DNA, RNA, peripheral blood mononuclear cells (PBMCs)

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or proven multiple sclerosis
* The participants are patients who are in inpatient or outpatient care of the Department of Neurology at the Medical University of Graz, Austria

Exclusion Criteria:

* Excluded from the examinations are all patients for whom an MRI examination is impossible or problematic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are patients who are in inpatient or outpatient care of the Department of Neurology at the Medical University of Graz, Austria with suspected or proven multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of EDSS ( Expanded Disability Status Scale) progression by combined markers of the disease | a maximum of 4 years
  EDSS score

SECONDARY OUTCOMES:
Prediction of clinical relapses | a maximum of 4 years
  Prediction of clinical relapses
Conversion from CIS (Clinically Isolated Syndrome) to MS (Multiple Sclerosis) defined by MRI and clinical criteria | a maximum of 4 years
  Conversion from CIS to MS defined by MRI and clinical criteria
Time of transition to progressive form of MS | a maximum of 4 years
  Time of transition to progressive form of MS
Neuropsychological progression (decrease in SDMT performance) | a maximum of 4 years
  Neuropsychological progression (decrease in SDMT performance)
Increase in morphological damage (lesion load, atrophy) | a maximum of 4 years
  Increase in morphological damage (lesion load, atrophy)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Enzinger, Prof, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided